CLINICAL TRIAL: NCT04679103
Title: A Safety and Immunogenicity Study in Long-term Treatment of Eculizumab (JSC "GENERIUM", Russian Federation) in Patients With Paroxysmal Nocturne Hemoglobinuria, Who Have Been Involved Earlier in the Clinical Trials of Eculizumab
Brief Title: A Safety and Immunogenicity Study in Long-term Treatment of Eculizumab (JSC "GENERIUM", Russian Federation)
Acronym: NAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECU-PNH-III-X; №205. eff.data 03 May 2018 (Other: Ministry of Health of the Russian Federation)
Record Dates: First submitted 2020-11-30; First posted 2020-12-22 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: eculizumab; humanized monoclonal antibodies; safety; paroxysmal nocturnal hemoglobinuria; rare disease; biosimilar; complement system; C5 component of complement; pro-inflammatory cytokines; Membrane attack complex (MAC); immunogenicity
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Rare Diseases | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: Interventional
Masking Description: NAP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculisumab (JSC GENERIUM, Russia) (Experimental): Eculizumab
  Interventions: Biological: Eculizumab (JSC GENERIUM, Russia)

INTERVENTIONS:
Biological: Eculizumab (JSC GENERIUM, Russia) — Eculizumab

SUMMARY:
A safety and immunogenicity study in long-term treatment of Eculizumab (JSC "GENERIUM", Russian Federation) in patients with paroxysmal nocturnal hemoglobinuria, who have been involved earlier in the clinical trials of Eculizumab (JSC "GENERIUM", Russian Federation).

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an ultra-rare, acquired, life-threatening, progressive clonal blood disease that is developed as a result of the expansion of one or more clones of hematopoietic stem cells with a somatic PIG A gene mutation. The main pathogenic mechanism of PNH development is a dysregulation of the complement system, in which there are no complement inhibitors CD55 and CD59 that are bounded by the GPI-anchor on the surface of blood cells, or there is a deficiency of them.

Eculizumab is the first drug for the pathogenetic therapy of PNH, a recombinant humanized monoclonal antibody against the C5 component of complement. Binding with high affinity to C5, eculizumab prevents the cleavage of C5 into C5a and C5b, thereby inhibiting the formation of pro-inflammatory cytokines (via C5a) and Membrane attack complex (MAC) (via C5b).

Using of eculizumab in patients with PNH leads to a significant decrease in hemolysis, the incidence of thrombosis and increasing of the quality of life of patients. It increases life expectancy with long-term using of eculizumab.

The drug Eculizumab, developed by JSC "GENERIUM", Russia, is a biological analogue (biosimilar) of the original drug Soliris®. At the present time Eculizumab (JSC GENERIUM, Russia) have already been authorized as Elizaria® in Russia.

This study is a multicenter open-label study of the safety, immunogenicity and efficacy of Eculizumab (JSC GENERIUM, Russia) in patients with paroxysmal nocturnal hemoglobinuria who completed participation in previous clinical trials of Eculizumab (JSC GENERIUM, Russia).

Visit 1 of this study is carried out on the day of the Visit of completion of a previously conducted study, or on another day, observing the terms of administration of the drug prescribed by the instructions for medical use of Eculizumab.

At this visit, all patients who signed the informed consent form and were immunized with meningococcal vaccine will begin therapy with Eculizumab (GENERIUM JSC), which will continue until the drug is registered or, as decided by the sponsoring company, until its commercial availability. When the last patient enrolled in the study has completed 6 months of therapy, which corresponds to the completion of Visit 13, an interim analysis of the safety and immunogenicity data of the study drug will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of participation in previous studies of Eculizumab (JSC "GENERIUM") while maintaining the clinical efficacy of the therapy with eculizumab.

   In case of significant deviations from the protocol during participation in previous studies, the decision on the possibility of patient participation in this study is made on an individual basis in agreement with the company Sponsor.
2. Written informed consent to participate in this study.
3. Documented vaccination against meningococcal infection (serotypes A, C, Y and W135 Neisseria meningitides) with an unexpired period of validity and consent of the patient to undergo booster vaccination against meningococcal infection (serotypes A, C, Y and W135 Neisseria meningitides) while participating in this research when the previous vaccination expires.
4. Consent to use a reliable method of contraception (a combination of at least 2 methods, including 1 barrier method, for example, using a condom and spermicide), from the moment of signing the informed consent until 10 weeks after the last administration of the study drug.

Exclusion Criteria:

1. Hypersensitivity to the study drug, as well as to its components.
2. Hypersensitivity to the active ingredients or any other component of the vaccine for the prevention of meningococcal infection, or a life-threatening reaction to the previous administration of a vaccine containing similar components.
3. Comorbidities and conditions that, in the opinion of the Investigator, endanger the safety of the patient while participating in the study.
4. Pregnancy or breastfeeding.
5. Alcohol, drug or drug addiction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of adverse events (AEs), serious adverse events (SAEs), including those associated with the use of the study drug. | 6 months
  Frequency of AE / SAE will be tabulated with an indication of the number and proportion of patients in each category. Data will be presented cumulatively for all patients, as well as by subgroup. Descriptive statistical methods will be used.
The number and proportion of patients with antidrug antibodies; titer of antidrug antibodies and their neutralizing activity. | 6 months
  The analysis of immunogenicity parameters will be carried out taking into account the total duration of treatment with eculizumab, including the results of previous studies. The baseline will be the results of the analysis before the first administration of the drug in clinical trials.If there is a sufficient number of data on the titer of antidrug antibodies and their neutralizing activity, they will be presented using descriptive statistics with additional indication of geometric means and coefficients of variation.
Changes in vital signs during the study. | 6 months
  Safety parameters, which are categorical variables (frequency of detection of abnormalities according to physical and instrumental examination data, the presence of abnormalities according to the results of ECG, Echo-CG and laboratory parameters) will be tabulated with an indication of number and proportion of patients in each category. Data will be presented cumulatively for all patients, as well as by subgroup.
Changes in physical examination during the study. | 6 months
  Safety parameters, which are categorical variables (frequency of detection of abnormalities according to physical and instrumental examination data, the presence of abnormalities according to the results of ECG, Echo-CG and laboratory parameters) will be tabulated with an indication of number and proportion of patients in each category. Data will be presented cumulatively for all patients, as well as by subgroup.
Changes in ECG during the study. | 6 months
  Safety parameters, which are categorical variables (frequency of detection of abnormalities according to physical and instrumental examination data, the presence of abnormalities according to the results of ECG, Echo-CG and laboratory parameters) will be tabulated with an indication of number and proportion of patients in each category. Data will be presented cumulatively for all patients, as well as by subgroup.
Changes in Doppler echocardiography during the study. | 6 months
  Safety parameters, which are categorical variables (frequency of detection of abnormalities according to physical and instrumental examination data, the presence of abnormalities according to the results of ECG, Echo-CG and laboratory parameters) will be tabulated with an indication of number and proportion of patients in each category. Data will be presented cumulatively for all patients, as well as by subgroup.

SECONDARY OUTCOMES:
Cmin will be carried out during the transition from the original Soliris® to the investigational drug. | 6 months
  The collection of blood samples will be carried out in patients who received Soliris® in the course of previous studies at Visits 1, 2, 3 and 4. 5-15 minutes before the start of the study drug administration.
The activity of the components of the complement system will be carried out during the transition from the original Soliris® to the investigational drug. | 6 months
  The collection of blood samples will be carried out in patients who received Soliris® in the course of previous studies at Visits 1, 2, 3 and 4. 5-15 minutes before the start of the study drug administration.
Concentration of membrane attack complex (C5b-9) will be carried out during the transition from the original Soliris® to the investigational drug. | 6 months
  The collection of blood samples will be carried out in patients who received Soliris® in the course of previous studies at Visits 1, 2, 3 and 4. 5-15 minutes before the start of the study drug administration.
Changes in LDH when switching from the original Soliris® to the investigational drug. | 6 months
  Methods of descriptive statistics will be used to analyze data on changes in laboratory parameters (LDH, hemoglobin, reticulocytes and creatinine) at various visits.
Changes in creatinine when switching from the original Soliris® to the investigational drug. | 6 months
  Methods of descriptive statistics will be used to analyze data on changes in laboratory parameters (LDH, hemoglobin, reticulocytes and creatinine) at various visits.
Changes in hemoglobin when switching from the original Soliris® to the investigational drug. | 6 months
  Methods of descriptive statistics will be used to analyze data on changes in laboratory parameters (LDH, hemoglobin, reticulocytes and creatinine) at various visits.
Changes in reticulocytes when switching from the original Soliris® to the investigational drug. | 6 months
  Methods of descriptive statistics will be used to analyze data on changes in laboratory parameters (LDH, hemoglobin, reticulocytes and creatinine) at various visits.
Changes in the size of PNH-clone of granulocytes and erythrocytes during the study. | 6 months
  Methods of descriptive statistics will be used to analyze data on changes in the size of PNH-clone of granulocytes and erythrocytes at various visits.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Markova, MD, Study Chair — AO GENERIUM
Locations (9):
- Russia (9):
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Chelyabinsk Oblast
  - Federal State Budgetary Institution of Science "Kirov Research Institute of Hematology and Blood Transfusion of the Federal Medical and Biological Agency", Kirov, Kirov Oblast
  - Federal State Budgetary Educational Institution of Higher Education "First St. Petersburg State Medical University named after Academician I.P. Pavlov", Saint Petersburg, Leningradskaya Oblast'
  - Federal State Budgetary Institution "National Medical Research Center of Hematology" of the Ministry of Health of the Russian Federation, Moscow, Moscow Oblast
  - State Budgetary Institution of Healthcare of the City of Moscow City Clinical Hospital named after S.P. Botkin of the Moscow Department of Health, Moscow, Moscow Oblast
  - State budgetary institution of health care of the Moscow region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow, Moscow Oblast
  - State budgetary institution of the Rostov region "Rostov Regional Clinical Hospital", Rostov-on-Don, Rostov Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara, Samara Oblast
  - State Budgetary Healthcare Institution of the Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No. 1", Yekaterinburg, Sverdlovsk Oblast

IPD SHARING:
Plan to Share IPD: No